CLINICAL TRIAL: NCT04413604
Title: Micronutrient Status in Children Aged 1-3 Years Consuming Their Habitual Diet With or Without Young Children's Milk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to recruitment difficulties
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19.08.INF
Record Dates: First submitted 2020-04-27; First posted 2020-06-04 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Nutritional Status; Child Nutrition Sciences

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YCM Group (1- <3) Years old (Experimental): 2 servings / day of the investigational (test) young children's milk (YCM) for 16 weeks
  Interventions: Other: Young children's milk (1-<3)
- Observation Group (1-<3) Years old (No Intervention): Habitual diet, consume the same regular foods and drinks as the children would normally

INTERVENTIONS:
Other: Young children's milk (1-<3) — young children's milk containing protein, energy and fat and micronutrients, in accordance with global and local nutritional recommendations for ages 1-3.
  Other Names: YCM
  Arms: YCM Group (1- <3) Years old

SUMMARY:
This study evaluates changes in Vitamin D, Zinc, and Iron status of children consuming 2 servings / day of the investigational (test) young children's milk (YCM) for 16 weeks compared to children of the same age who consume their habitual pattern of beverage intake for the same duration.

DETAILED DESCRIPTION:
The overall purpose of the study is to demonstrate improved vitamin D status and/or improved iron status of children ages 1 to 3 years who are consuming the investigational (test) young children's milk (YCM) compared to children consuming their habitual pattern of beverage intake (milk and non-milk beverages). This is based on previous study findings that (i) the toddler's diet, in reality, is often not optimal, putting toddlers at risk of insufficient intakes of several nutrients, and (ii) consuming YCM supplemented with these nutrients might provide optimal intakes of these nutrients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained from the parent.
* Full-term gestational birth (≥ 37 completed weeks of gestation), with a birth weight of ≥ 2.5 kg and ≤ 4.5 kg.
* Child is age 12 - 32 months at enrolment.
* Child is no longer being breastfed (neither exclusively nor partially)
* Child's parent is of legal age of consent, must understand the informed consent form and other study documents, and is willing and able to fulfill the requirements of the study protocol.

Exclusion Criteria:

* Child has consumed micronutrient supplements or micronutrient fortified foods or beverages in amounts greater than the thresholds below:

  1. Micronutrient supplements (except for vitamin A): zero in the past 4 weeks
  2. Micronutrient-fortified foods or beverages: zero servings in the past 2 weeks
* Chronic infectious illness, helminthiasis, or other acute disease/disorder potentially affecting feeding or growth (mild infectious illness, such as acute viral rhinopharyngitis, is acceptable).
* Any congenital malformation (e.g., gastrointestinal tract atresia) or surgery sequelae (e.g. short bowel syndrome) potentially affecting feeding, growth, or nutrient absorption.
* Child exhibits any clinical signs of potential micronutrient deficiencies (e.g., hemoglobin < 100 g/L based on screening assessment, rickets based on physical exam).
* Known or suspected cows' milk protein intolerance / allergy, lactose intolerance, soy intolerance / allergy, fish oil intolerance / allergy, or other food allergies that affect diet.
* Child fed vegan, vegetarian, or vegetarian plus fish diets in which milk products are excluded.
* Weight-for-age value < -2 or > 2 standard deviations from the WHO(world health organization) Child Growth Standards median at enrollment.
* Height-for-age < -2 or > 2 standard deviations from the WHO(world health organization) Child Growth Standards median at enrollment.
* Child has participated in another clinical trial within 4 weeks prior to enrollment.
* Child of any investigational site staff member or Nestle employee directly involved in the conduct of the trial.
* Other medical or psychiatric condition that, in the judgement of the investigator, would make the child inappropriate for entry into the study.

Ages: 12 Months to 32 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
change in Vitamin D and Iron status | 16 weeks
  measure blood vitamin D and Iron value

SECONDARY OUTCOMES:
change in Zinc status | 16 weeks
  measure blood Zinc value
Assess micronutrient intake | 16 weeks
  Using 24 hour dietary recall

OTHER OUTCOMES:
assess other nutrient biomarkers | 16 weeks
  measure changes by blood measurement for CRP in mg/L
assess other nutrient biomarkers | 16 weeks
  measure changes by blood measurement for serum retinol in μmol/L
assess other nutrient biomarkers | 16 weeks
  measure changes by blood measurement for alpha(1)-acid glycoprotein in absolute value
assess muscular fitness | 16 weeks
  measure changes by blood measurement for serum niacin
assess muscular fitness | 16 weeks
  measure changes by blood measurement for plasma vitamin B6
assess child developmental milestones | 16 weeks
  measure Ages & Stages Questionnaires, Third Edition; Minimum 0, Maximum 60, higher scores indicate more positive outcomes
assess child developmental milestones | 16 weeks
  measure Ages & Stages Questionnaires: Social-Emotional, Second Edition, Minimum 0, Maximum 180, lower scores indicate more positive outcomes
assess bone mass index | 16 weeks
  measure the development of bone mass
assess muscular fitness | 16 weeks
  measure handgrip strength using a portable dynamometer
assess stool microbiota composition and metabolism and gut biomarkers | 16 weeks
  measure stool microbiota composition and metabolism, plus biomarkers of gut function (e.g., calprotectin, alpha-1 antitrypsin, albumin) and short-chain fatty acids.
assess genetic markers of vitamin D metabolism / status | baseline
  measure genetic variants isolated from blood draw
assess gastrointestinal (GI) tolerance | 16 weeks
  measure changes in gut comfort level min 10, max 60. Lower score indicate more positive outcomes
assess YCM acceptability in children consuming GUM. | 16 weeks
  measure how well acceptable is YCM for interventional group, minimum score 5 max score 33. higher score indicate positive outcome
To monitor growth and development | 16 weeks
  Anthropometry Assessment based on BMI in (kg/m^2) by weight (Kilograms), height (Metres)
To monitor standard adverse events (AE) | 16 weeks
  safety assessment by monitoring the AEs linked with participation in study
To monitor absenteeism from day care or pre-school due to illness | 16 weeks
  safety assessment by monitoring the days of absenteeism linked with participation in study
To monitor concomitant medication (CM) reporting | 16 weeks
  safety assessment by monitoring the concomitant medication linked with participation in study

CONTACTS AND LOCATIONS:
Overall Officials: Sudigdo Sastroasmoro, MD, Principal Investigator — Department of Child Health, Medical School, University of Indonesia
Locations (1):
- Indonesian Nutrition Association, Jakarta Pusat, Jakarta Special Capital Region, Indonesia